CLINICAL TRIAL: NCT03500991
Title: Phase 1 Study of HER2-Specific CAR T Cell Locoregional Immunotherapy for HER2 Positive Recurrent/Refractory Pediatric Central Nervous System Tumors
Brief Title: HER2-specific CAR T Cell Locoregional Immunotherapy for HER2-positive Recurrent/Refractory Pediatric CNS Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Immunotherapy, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrainChild-01
Record Dates: First submitted 2018-03-21; First posted 2018-04-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Tumor, Pediatric; Glioma; Ependymoma; Medulloblastoma; Germ Cell Tumor; Atypical Teratoid/Rhabdoid Tumor; Primitive Neuroectodermal Tumor; Choroid Plexus Carcinoma; Pineoblastoma
Keywords: CNS, CAR T cell, HER2-positive, brain tumor; pediatric, young adults
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Ependymoma; Medulloblastoma; Neoplasms, Germ Cell and Embryonal; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Choroid Plexus Carcinoma; Pinealoma; Brain Neoplasms | interventions — Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM A (Tumor Cavity Infusion) (Experimental): patients with supratentorial tumors for which CAR T cells will be delivered into the tumor resection cavity
  Intervention: HER2-specific chimeric antigen receptor (CAR) T cell
  Interventions: Biological: HER2-specific chimeric antigen receptor (CAR) T cell
- ARM B (Ventricular System Infusion) (Experimental): patients with either infratentorial tumors or leptomeningeal tumors for which the CAR T cells will be delivered into the fourth ventricle or lateral ventricle, respectively
  Intervention: HER2-specific chimeric antigen receptor (CAR) T cell
  Interventions: Biological: HER2-specific chimeric antigen receptor (CAR) T cell

INTERVENTIONS:
Biological: HER2-specific chimeric antigen receptor (CAR) T cell — Autologous CD4 and CD8 T cells lentivirally transduced to express a HER2 specific chimeric antigen receptor (CAR) and EGFRt given via indwelling central nervous system (CNS) catheter

SUMMARY:
This is a Phase 1 study of central nervous system (CNS) locoregional adoptive therapy with autologous CD4 and CD8 T cells lentivirally transduced to express a HER2-specific chimeric antigen receptor (CAR) and EGFRt, delivered by an indwelling catheter in the tumor resection cavity or ventricular system in children and young adults with recurrent or refractory HER2-positive CNS tumors. A child or young adult with a refractory or recurrent CNS tumor will have their tumor tested for HER2 expression by immunohistochemistry (IHC) at their home institution or at Seattle Children's Hospital. If the tumor is HER2 positive and the patient meets all other eligibility criteria, including having a CNS catheter placed into the tumor resection cavity or into their ventricular system, and meets none of the exclusion criteria, then they can be apheresed, meaning T cells will be collected. The T cells will then be bioengineered into a second-generation CAR T cell that targets HER2-expressing tumor cells. The patient's newly engineered T cells will then be administered via the indwelling CNS catheter for two courses. In the first course they will receive a weekly dose of CAR T cells for three weeks, followed by a week off, an examination period, and then another course of weekly doses for three weeks. Following the two courses, patient's will undergo a series of studies including MRI to evaluate the effect of the CAR T cells and may have the opportunity to continue receiving additional courses of CAR T cells if the patient has not had adverse effects and if more of their T cells are available.

The hypothesis is that an adequate amount of HER2-specific CAR T cells can be manufactured to complete two courses of treatment with three doses given on a weekly schedule followed by one week off in each course. The other hypothesis is that HER-specific CAR T cells safely can be administered through an indwelling CNS catheter to allow the T cells to directly interact with the tumor cells for each patient enrolled on the study safely can be delivered directly into the brain via indwelling catheter. Secondary aims of the study will include to evaluate CAR T cell distribution with the cerebrospinal fluid (CSF), the extent to which CAR T cells egress or traffic into the peripheral circulation or blood stream, and, if tissues samples from multiple time points are available, also evaluate the degree of HER2 expression at diagnosis versus at recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 and ≤ 26 years
2. Histologically diagnosed HER2-positive Central Nervous System (CNS) tumor
3. Evidence of refractory or recurrent CNS disease for which there is no standard therapy
4. Able to tolerate apheresis, or has apheresis product available for use in manufacturing
5. CNS reservoir catheter, such as an Ommaya or Rickham catheter
6. Life expectancy ≥ 8 weeks
7. Lansky or Karnofsky score ≥ 60
8. If patient does not have previously obtained apheresis product, patient must have recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy and discontinue the following prior to enrollment:

   1. ≥ 7 days post last chemotherapy/biologic administration
   2. 3 half-lives or 30 days, whichever is shorter post last dose of anti-tumor antibody therapy
   3. Must be at least 30 days from most recent cell infusion
   4. All systemically administered corticosteroid treatment therapy must be stable or decreasing within 1 week prior to enrollment with maximum dexamethasone dose of 2.5 mg/m2/day. Corticosteroid physiologic replacement therapy is allowed.
9. Adequate organ function
10. Adequate laboratory values
11. Patients of childbearing/fathering potential must agree to use highly effective contraception

Exclusion Criteria:

1. Diagnosis of classic diffuse intrinsic pontine glioma (DIPG)
2. Presence of Grade ≥ 3 cardiac dysfunction or symptomatic arrhythmia requiring intervention
3. Presence of primary immunodeficiency/bone marrow failure syndrome
4. Presence of clinical and/or radiographic evidence of impending herniation
5. Presence of active malignancy other than the primary CNS tumor under study
6. Presence of active severe infection
7. Pregnant or breastfeeding
8. Subject and/or authorized legal representative unwilling or unable to provide consent/assent for participation in the 15-year follow up period
9. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2039-07-26 (Estimated)

PRIMARY OUTCOMES:
Establish the safety, defined by the adverse events, of HER2-specific CAR T cell infusions delivered by a central nervous system (CNS) catheter into the tumor resection cavity or ventricular system | up to 6 months
  The type, frequency, severity, and duration of adverse events as a result of HER2-specific CAR T cell infusion will be summarized
Establish the feasibility, defined by the ability to produce and administer CAR T cell product, of HER2-specific CAR T cell product infusions delivered by a central nervous system (CNS) catheter into the tumor resection cavity or ventricular system | 28 days
  The proportion of products successfully manufactured and infused will be measured

SECONDARY OUTCOMES:
Assess the distribution of CNS-delivered HER2-specific CAR T cells within the cerebrospinal fluid (CSF) and peripheral blood | up to 6 months
  The trafficking of HER2-specific CAR T cell product through the CSF by measuring remaining CAR T cells from a prior infusion at the time of each infusion and the trafficking of HER2-specific CAR T cells from the CSF into the peripheral blood will be evaluated
Assessment of whether HER2 expression changes in relapsed CNS tumors that were HER2 positive prior to treatment with CAR T cells | 28 days
  The changes in HER2 expression at diagnosis and recurrence of central nervous system (CNS) tumors, if samples from multiple time points is available, will be investigated by evaluating pathology specimens from previous surgeries
Assessment of disease response of HER2-expressing refractory or recurrent central nervous system (CNS) tumors to HER2 specific CAR T cell therapy delivered directly into the CNS | up to 6 months
  The response of recurrent or refractory central HER2-expressing CNS tumors to HER2-specific CAR T cell therapy delivered directly into the CNS will be determined by evaluating CSF for tumor cells and by CNS imaging with MRIs

OTHER OUTCOMES:
Analysis of CSF for biomarkers of anti-tumor CAR T cell functional activity | up to 6 months
  The presence of biomarkers of CAR T cell functional activity, such as cytokines, will be quantified via protein expression analysis in CSF. These findings will be correlated with safety determined by occurrence of adverse events, and response determined by disease evaluations via CSF cytology and MRI imaging of the CNS.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ronsley, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Li W, Xu L, Song Y. Chimeric antigen receptor-immune cells against solid tumors: Structures, mechanisms, recent advances, and future developments. Chin Med J (Engl). 2024 Jun 5;137(11):1285-1302. doi: 10.1097/CM9.0000000000002818. Epub 2023 Aug 28. PMID 37640679
- [Derived] Vitanza NA, Johnson AJ, Wilson AL, Brown C, Yokoyama JK, Kunkele A, Chang CA, Rawlings-Rhea S, Huang W, Seidel K, Albert CM, Pinto N, Gust J, Finn LS, Ojemann JG, Wright J, Orentas RJ, Baldwin M, Gardner RA, Jensen MC, Park JR. Locoregional infusion of HER2-specific CAR T cells in children and young adults with recurrent or refractory CNS tumors: an interim analysis. Nat Med. 2021 Sep;27(9):1544-1552. doi: 10.1038/s41591-021-01404-8. Epub 2021 Jul 12. PMID 34253928